CLINICAL TRIAL: NCT05248373
Title: A Randomized Double-blind Placebo-controlled Multi-center Clinical Trial in Parallel Assignment of Safety, Tolerability and Immunogenicity of a Vaccine "Gam-COVID-Vac, a Combined Vector Vaccine for the Prevention of Coronavirus Infection Caused by the SARS-CoV-2 Virus" in a Nasal Spray Dosage Form With the Participation of Adult Volunteers
Brief Title: Safety, Tolerability and Immunogenicity of Gam-COVID-Vac Vaccine in a Nasal Spray
Acronym: SPRAY
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SPRAY vaccine against COVID-19
Record Dates: First submitted 2022-02-07; First posted 2022-02-21 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; SARS-CoV-2 Acute Respiratory Disease
Keywords: vaccine; Sputnik; adenoviral vector vaccine; intranasal vaccine
MeSH Terms: conditions — COVID-19 | interventions — Gam-COVID-Vac vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rAd26 single administration (Experimental)
  Interventions: Biological: Gam-COVID-Vac
- rAd5 single administration (Experimental)
  Interventions: Biological: Gam-COVID-Vac
- prime-boost regimen with rAd26 followed rAd5 administration (Experimental)
  Interventions: Biological: Gam-COVID-Vac
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Gam-COVID-Vac — two-component combined vector vaccine for the prevention of coronavirus infection caused by the SARS-CoV-2 virus
  Arms: prime-boost regimen with rAd26 followed rAd5 administration; rAd26 single administration; rAd5 single administration
Other: Placebo — solution with same composition as for vaccine formulation except rAds
  Arms: placebo

SUMMARY:
Randomized, double-blind, placebo-controlled trial to evaluate safety and immunogenicity of intranasal "Gam-COVID-Vak" combined vector vaccine for the prevention of coronavirus infection caused by the SARS-CoV-2 virus.

The duration of participation in the study for one subject will be 180±14 days after the first dose of vaccine, during which each subject will undergo a screening visit (within a week) and face-to-face visits according to the study plan. Intranasal vaccine administration will be done at day 1 vaccination visits and day 21±2 days on an outpatient basis.

During the follow-up visits key vital signs will be assessed, and will collect data on changes in the state and well-being subjects from a previous visit. Subject data will be collected using electronic forms of individual registration cards, as well as with using questionnaires (diaries) filled by the subjects of the study.

Immunogenicity will be assessed on day 1, 10, 28, 42 and 90 days. Humoral and cellular immune response will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of a written informed consent of the subject to participate in the study;
2. Adult volunteers over 18;
3. Negative test result for HIV, hepatitis, syphilis;
4. Negative test result for COVID-2019, determined by PCR at the visit screening, and, if available, the result of the examination performed in medical organizations that are research centers 7 days before inclusion into research;
5. The result of the study for the presence of IgG antibodies to SARS CoV2 up to 10 VGR, which corresponds to value up to 100 BAU, regardless of the immune status before;
6. Absence of contact of the research subject with patients with COVID-2019 for at least 14 days before enrollment in the study (according to the study participant);
7. Consent to use effective methods of contraception during the entire period of participation in research;
8. Negative Urine Pregnancy Test at Screening Visit (for women of childbearing age);
9. Negative test for the presence of narcotic and psychostimulant drugs in the urine for screening visit;
10. Negative alcohol test at screening visit;
11. No history of severe post-vaccination reactions or post-vaccination complications after the use of immunobiological preparations;
12. Absence of acute infectious and/or respiratory diseases for at least within 14 days prior to enrollment in the study.

Exclusion Criteria:

1. Inability to give informed consent, inability to understand the essence of the study
2. Any vaccination/immunization carried out within 30 days prior to inclusion in study;
3. Steroid therapy (excluding hormonal contraceptives) and/or immunoglobulins or other blood products, not completed 30 days before inclusion in the study;
4. COVID-2019 disease or vaccination to prevent COVID-2019 in less than six months before inclusion in the study
5. Immunosuppressive drug therapy completed less than 3 months before inclusion in the study;
6. Postponed less than one year prior to enrollment in the study acute coronary syndrome or stroke;
7. Tuberculosis, chronic systemic infections;
8. Exacerbation of rhinitis
9. Burdened allergic history (presence in the anamnesis of information about anaphylactic shock, angioedema, polymorphic exudative eczema, serum sickness), hypersensitivity or allergic reactions to the introduction of immunobiological drugs, known allergic reactions to drug components, exacerbation allergic diseases on the day of inclusion in the study;
10. History of neoplasms (ICD codes C00-D09);
11. Donation of blood or plasma (in a volume of 450 ml or more) less than 2 months before inclusion in the study;
12. Splenectomy in history;
13. Neutropenia (decrease in the absolute number of neutrophils less than 1000/mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin less than 80 g/l), immunodeficiency in history within 6 months prior to enrollment in the study;
14. Subjects with active human immunodeficiency virus disease syphilis, hepatitis B and C;
15. Anorexia, protein deficiency of any origin;
16. History of alcoholism and drug addiction;
17. Participation of the subject in any other interventional clinical trial during this study;
18. Any other condition of the research subject that, in the opinion of the research physician, may prevent completion of the study in accordance with the protocol;
19. Staff of research centers and other staff directly involved in conducting the study (principal investigator and members of the research team) and members of their families.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-03-08 (Estimated); Primary Completion 2023-02-14 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in geometric mean titer of IgGs specific to S protein | 0, 10, 28, 42, 90 day
  Change from baseline in Geometric mean titer of IgGs specific to S protein at different time points after vaccination
Change from baseline in number of participants with detected specific IgGs | 0, 10, 28, 42, 90 day
  Change from baseline in Number of participants with detected specific IgGs at different time points after vaccination
Change from baseline in Number of participants with detected specific IgAs | 0, 10, 28, 42 day
  Change from baseline in Number of participants with detected specific IgAs at different time points after vaccination
Change from baseline in Geometric mean titer of neutralizing antibodies to SARS-Cov-2 virus | 0, 28, 42, 90 day
  Change from baseline in Geometric mean titer of neutralizing antibodies to SARS-Cov-2 virus at different time points after vaccination
Change from baseline in Number of participants with detected neutralizing antibodies to SARS-Cov-2 virus | 0, 28, 42, 90 day
  Change from baseline in Number of participants with detected neutralizing antibodies to SARS-Cov-2 virus at different time points after vaccination
Proportion of participants with any adverse events | 1-180 days
  AEs evaluation during the whole period of the study
Proportion of participants with severe adverse events | 1-180 days
  SAEs evaluation during the whole period of the study

SECONDARY OUTCOMES:
Efficacy of symptomatic COVID-19 prevention | 28-180 days
  Efficacy of symptomatic COVID-19 prevention

IPD SHARING:
Plan to Share IPD: No